CLINICAL TRIAL: NCT05309694
Title: A Post-Marketing, Prospective, Multi-Center, Single Arm, Open Label Clinical Study to Evaluate the Safety of a New Inserter Design for Paragard® T380A Intrauterine Copper Contraceptive
Brief Title: A Study to Assess the Safety of a New Inserter Device for Paragard® (Intrauterine Copper Contraceptive)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CooperSurgical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CSIPD-001
Record Dates: First submitted 2022-03-07; First posted 2022-04-04 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Contraception
Keywords: Contraception; Copper Intrauterine Device; Intrauterine Device; Contraceptive; Birth Control; IUD; IUS; Intrauterine System

STUDY DESIGN:
Intervention Model Description: Single arm and open-label design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Group 1 (Other): Paragard® T380A Intrauterine Copper Contraceptive with new inserter Non parous and parous female subjects of child bearing potential
  Interventions: Combination Product: Paragard® T380A Intrauterine Copper Contraceptive with New Inserter

INTERVENTIONS:
Combination Product: Paragard® T380A Intrauterine Copper Contraceptive with New Inserter — Paragard® IUS with Investigational Inserter combines the current insertion tube and white rod to form a new pre-assembled inserter device that supports a single hand operation.
  The device is used to pass the IUS through the cervical canal and into the uterine cavity and facilitates insertion of the T shaped Paragard® IUS implant into the uterus.

SUMMARY:
The purpose of this study is to demonstrate that a new device inserter leads to successful and safe insertion of Paragard® IUS, comparable to the currently approved IUS inserter, in females of reproductive potential.

DETAILED DESCRIPTION:
This is a post-market prospective clinical study to be conducted at multiple centers in a single arm and open-label design to evaluate the safety of a new inserter design for Paragard® (intrauterine copper contraceptive). The study will be conducted in female subjects of child bearing potential.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a postmenarcheal and premenopausal woman of child bearing potential.
* Subjects are at least 18 years of age, at the time of signing the informed consent.
* Subject is overtly healthy as determined by medical evaluation.

Exclusion Criteria:

* Pregnancy or suspicion of pregnancy or at risk for luteal phase pregnancy
* History of previous IUD complications
* Abnormalities of the uterus resulting in distortion of the uterine cavity that may complicate IUD insertion
* Known anatomical abnormalities of the cervix
* Presence of acute pelvic inflammatory disease at the time of screening.
* Postpartum endometritis.
* Known or suspected uterine or cervical malignancy.
* Uterine bleeding of unknown etiology.
* Untreated acute cervicitis or vaginitis or other lower genital tract infection.
* Conditions associated with increased susceptibility to pelvic infections.
* Subjects with Wilson's disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Successful Insertions | From enrollment to end of treatment at 3 months
  The percentage of successful insertions will be calculated by number of subjects with successful insertions relative to the total number of subjects with at least one successful or unsuccessful insertion attempt.

SECONDARY OUTCOMES:
Uterine Perforation and IUD Embedment | From enrollment to end of treatment at 3 months
  Frequency of uterine perforation and IUD embedment
IUS Expulsions and Dislocations | From enrollment to end of treatment at 3 months
  Frequency of IUS expulsions (partial or total) and dislocations
Adverse Events | From enrollment to end of treatment at 3 months
  Frequency of Serious Adverse Events (SAE) and Adverse Events (AE)
Adverse Events related to Procedure | From enrollment to end of treatment at 3 months
  Frequency of AEs related to procedure
Vasovagal Events | From enrollment to end of treatment at 3 months
  Frequency of vasovagal events at the time of insertion
Pelvic Infections | From enrollment to end of treatment at 3 months
  Frequency of pelvic infections related to IUS insertion and use

CONTACTS AND LOCATIONS:
Overall Officials: Robin Kroll, MD, Principal Investigator — Seattle Clinical Research Center; Carol Stamm, MD, Principal Investigator — Downtown Women's Healthcare; Joyce Miller, MD, Principal Investigator — South Miami Women's Health; Jacquelyn Robinson, MD, Principal Investigator — Valley Ob-Gyn Clinic, PC; Ronald Hirth, MD, Principal Investigator — Hilltop Obstetrics & Gynecology; Mark Akin, MD, Principal Investigator — Austin Area Ob-Gyn & Fertility; Stephanie Reich, MD, Principal Investigator — Central Austin - Women Partners in Health; Eric L Brown, MD, Principal Investigator — GYN-CARE Women's Healthcare
Locations (8):
- United States (8):
  - Downtown Women's Healthcare, Denver, Colorado
  - South Miami Women's Health, South Miami, Florida
  - GYN-CARE Women's Healthcare, Atlanta, Georgia
  - Valley Ob-Gyn Clinic, PC, Saginaw, Michigan
  - Hilltop Obstetrics & Gynecology, Franklin, Ohio
  - Central Austin - Women Partners in Health, Austin, Texas
  - Austin Area Ob-Gyn & Fertility, Austin, Texas
  - Seattle Clinical Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dunsmoor-Su RF, Desai VB, Pandolfi EC, Audette CR, Miller JR, Fuller AE, Brown EL, Hirth RD, Seetal-Kihei KV, McKain LF. Placement of the T380A Intrauterine Copper Contraceptive Using a Single-Hand Inserter. O G Open. 2025 Mar 6;2(2):e068. doi: 10.1097/og9.0000000000000068. eCollection 2025 Apr. PMID 41000288